CLINICAL TRIAL: NCT03550755
Title: Open Label Single Arm Phase II Immunotherapy Trial in Patients With Cervical Cancer
Brief Title: Immunotherapy of Cervical Cancer With V3-Cervix
Acronym: V3-Cervix
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V3-Cervix-01
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Cervical Cancer
Keywords: cervix; uterus
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group assignment to receive one pill of vaccine once per day for 3 months
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V3-Cervix (Experimental): Biological: V3-Cervix V3-Cervix is a tableted immunotherapeutic derived from hydrolyzed, heat-inactivated, pooled blood and tumor tissue from women with cervical cancer
  Interventions: Biological: V3-Cervix

INTERVENTIONS:
Biological: V3-Cervix — Oral tableted preparation containing hydrolyzed tumor antigens derived from peripheral blood and tumor tissue

SUMMARY:
The goal of this trial is to evaluate the efficacy of immunotherapy for cervical cancer based on a fundamentally new approach. We will test new tableted preparation, V3-Cervix, obtained from hydrolyzed, inactivated blood and tumors of patients with cervical cancer. When administered orally, it should cause a specific anti-tumor immune response and an anti-inflammatory effect. Trial is planned to last 3 months, recruit 20 volunteers, administer daily pill of vaccine and evaluate effect on tumor size and tumor markers.

DETAILED DESCRIPTION:
Cervical cancer (CC) is a malignant neoplasm that occurs in the cervix. Histologically, there are two main types: adenocarcinoma and squamous cell carcinoma. Cervical cancer is most common in middle-aged women (35-55 years of age), in 20% of cases it is found over the age of 65 years. Cancer of the body and cervix are the most common type of malignant tumor of female genital organs. It is believed that human papillomavirus (HPV) is the main risk factor causing cervical cancer. Cervical cancer combines surgical treatment, radiotherapy and chemotherapy. Current immunotherapies did not show much success. The prognosis depends on the stage of the disease: 5-year survival rate at the first stage is 78.1%, at the second stage - 57%, at the third - 31%, at the fourth - 7.8%. There is no specific cervical cancer marker, usually a panel of markers is used including CA125, beta-hCG, CEA, SCC, CA19.9 and CA27.29. The goal of this trial is to evaluate the efficacy of immunotherapy for cervical cancer based on a fundamentally new approach. We will test new tableted preparation, V3-Cervix, obtained from hydrolyzed, inactivated blood and tumors of patients with cervical cancer. When administered orally, it should cause a specific anti-tumor immune response and an anti-inflammatory effect. Trial is planned to last 3 months, recruit 20 volunteers, administer daily pill of vaccine and evaluate effect on tumor size and tumor markers.

ELIGIBILITY:
Inclusion Criteria:

confirmed diagnosis of cervical cancer available baseline measurement of tumor size and burden presence of tumor markers associated with cervical cancer, i.e., CA125, beta-hCG, CEA, SCC, СА19.9 and СА27.29 -

Exclusion Criteria:

metastases to other sites hysterectomy

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This particular condition, i.e., cervical cancer, is gender specific as it is found in females only
Enrollment: 20 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in tumor size and burden compared to baseline | monthly for 3 months
  Intravaginal ultrasonography of lower abdomen to measure changes

SECONDARY OUTCOMES:
Effect on baseline tumor markers, if any | Monthly for three months
  Change in serum levels of a panel of tumor markers such as CA125, beta-hCG, CEA, SCC, СА19.9 and СА27.29 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbaiar, PhD, MD/PhD, Study Chair — Immunitor Inc.
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No
Data will be available upon study conclusion